CLINICAL TRIAL: NCT02159690
Title: A Phase II Neoadjuvant Study of Enzalutamide, Abiraterone Acetate, Dutasteride and Degarelix in Men With Localized Prostate Cancer Pre-prostatectomy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of funding
Sponsor: Kenneth Pienta, MD (Other)
Collaborators: Prostate Cancer Foundation Norway (Unknown)
Responsible Party: Sponsor-Investigator, Kenneth Pienta, MD, Principal Investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neoadj enz/abi/dut/deg
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer; Localized Prostate Cancer
Keywords: prostate cancer; prostatectomy; localized prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Abiraterone Acetate; Prednisone; Dutasteride; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

INTERVENTIONS:
Drug: Enzalutamide — 160mg
  Other Names: MDV3100; Xtandi
Drug: Abiraterone acetate — 1000mg
  Other Names: Zytiga
Drug: Prednisone — 5mg twice daily (to blunt mineralocorticoid side effects from abiraterone)
  Other Names: Deltasone
Drug: Dutasteride — 0.5mg
  Other Names: Avodart
Drug: Degarelix — 240mg SC loading dose on day 1, then three 80mg SC injections every 4 weeks thereafter
  Other Names: Firmagon

SUMMARY:
This study investigates the pathologic effects of the combination of enzalutamide, abiraterone acetate, dutasteride, and degarelix when given for 12 weeks prior to prostatectomy in men with localized prostate cancer.

Enzalutamide, an androgen receptor (AR) antagonist, blocks binding of testosterone to the AR as well as preventing nuclear translocation of the AR and DNA binding. Abiraterone acetate inhibits the CYP17 pathway, which is involved in the formation of androgens. Dutasteride is a 5-alpha-reductase inhibitor which blocks conversion of testosterone to dihydrotestosterone. Degarelix, a gonadotropin-releasing hormone (GnRH) antagonist, binds to GnRH receptors on the pituitary gland thus suppressing testosterone release from the testes.

Therefore it is hypothesized that the combination of enzalutamide, abiraterone acetate, dutasteride, and degarelix will result in near-complete AR inhibition and produce favorable pathologic changes after 12 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 years
3. Eastern cooperative group (ECOG) performance status ≤2
4. Documented histologically confirmed adenocarcinoma of the prostate
5. Willing to undergo prostatectomy as primary treatment for localized prostate cancer
6. High risk prostate cancer (per NCCN criteria): Gleason score 8-10 or T3a or PSA > 20 ng/mL -Or- Very-high risk prostate cancer (per NCCN criteria): T3b -T4
7. Serum testosterone ≥150 ng/dL
8. Able to swallow the study drugs whole as tablets
9. Willing to take abiraterone acetate on an empty stomach (no food should be consumed at least two hours before and for one hour after dosing).
10. Willing to use a condom if having sex with a pregnant woman, or use a condom and another effective method of birth control if having sex with a woman of child-bearing potential. These measures are required during and for one week after treatment with abiraterone.

Exclusion Criteria:

1. Prior local therapy to treat prostate cancer (e.g. radical prostatectomy, radiation therapy, brachytherapy)
2. Prior use of enzalutamide or abiraterone acetate
3. Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

   1. Hormonal therapy (e.g. leuprolide, goserelin, triptorelin, degarelix)
   2. CYP-17 inhibitors (e.g. ketoconazole)
   3. Antiandrogens (e.g. bicalutamide, nilutamide)
   4. Second generation antiandrogens (e.g. enzalutamide, ARN-509)
   5. Immunotherapy (e.g. sipuleucel-T, ipilimumab)
   6. Chemotherapy (e.g. docetaxel, cabazitaxel)
4. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
5. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
6. Abnormal bone marrow function [absolute neutrophil count (ANC)<1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL]
7. Abnormal liver function (bilirubin, AST, ALT ≥ 3 x upper limit of normal)
8. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
9. Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within the last five years prior to enrollment in the study.
10. History of prior cardiac arrhythmia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of prostatectomy specimens with a complete response rate | 12 weeks
  Proportion of prostatectomy specimens with complete response rate after 12 weeks of therapy

SECONDARY OUTCOMES:
Proportion of prostatectomy specimens with a negative surgical margin rate | 12 weeks
  Proportion of prostatectomy specimens with a negative surgical margin rate after 12 weeks of therapy
Proportion of prostatectomy specimens with a near-pathologic complete response | 12 weeks
  Proportion of prostatectomy specimens with a near-pathologic complete response (<=5mm of residual tumor) after 12 weeks of therapy
Proportion of prostatectomy specimens with pathologic T3 disease | 12 weeks
  Proportion of prostatectomy specimens with pathologic T3 disease after 12 weeks of therapy
Change in immunologic parameters (TREC levels and antibody responses) | 16 weeks
  Change in immunologic parameters (TREC levels and antibody responses) after 12 weeks of enzalutamide, abiraterone acetate, dutasteride and degarelix and an additional month of degarelix monotherapy (16 weeks total).
Proportion of radiographic disappearance of MRI detectable significant prostate nodules | 12 weeks
  Proportion of radiographic disappearance of MRI detectable significant prostate nodules after 12 weeks of therapy.
Proportion of men who receive adjuvant radiation therapy within 1 year of prostatectomy | 64 weeks
  Proportion of men who receive adjuvant radiation therapy within 1 year of prostatectomy (12 weeks of therapy + 1 year = 64 weeks)
PSA progression free survival | 2 years after last accrual
  The biochemical (i.e. PSA) progression free survival estimate two years after the last patient has accrued.
Overall survival | 2 years after last accrual
  The overall survival estimate two years after the last patient has accrued.
Incidence and severity of adverse events | 16 weeks
  Safety as assessed by the incidence and severity of adverse events and serious adverse events graded according to the National Cancer Institute - Common Terminology Criteria for adverse events (CTCAE) version 4.0
Exploratory biomarkers assessment | 16 weeks
  Exploratory biomarker Assessment. Examples of these may include, but are not limited to: assessment for genomic PTEN loss via fluorescence in situ hybridization (FISH), PTEN immunohistochemistry (IHC), assessment for alteration in MYC/chromosome 8q24 via FISH, RNAseq analysis, serum drug/androgen levels and intraprostatic drug/androgen levels.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Pienta, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States